CLINICAL TRIAL: NCT01329666
Title: Early Effect of Vitamin D in Primary Hyperparathyroidism
Brief Title: Primary Hyperparathyroidism (PHPT): Early Effect of Vitamin D
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shonni J. Silverberg, Professor of Medicine, Endocrinology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AAAF1846; R01DK084986 (NIH)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Primary Hyperparathyroidism; Hypercalcemia; Vitamin D Deficiency; Osteoporosis; Osteopenia
Keywords: Primary Hyperparathyroidism; Endocrinology; Hypercalcemia; Vitamin D deficiency; Parathyroid Hormone; Osteoporosis; Bone Density; Vitamin D repletion; Vitamin D Supplements
MeSH Terms: conditions — Hyperparathyroidism, Primary; Hypercalcemia; Vitamin D Deficiency; Osteoporosis; Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 50,000 IU Vitamin D3 (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (inactive Vitamin D3) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects will receive placebo vitamin D3, 1 pill weekly for 12 weeks.
  Arms: Placebo (inactive Vitamin D3)
Dietary Supplement: Vitamin D3 — Baseline:
  50,000 IU/week for 8 weeks
  Week 8:
  Subjects with D3 less than 30 ng/ml: 50,000 IU/week for 4 weeks.
  Subjects with D3 25-OHD at or above 30 ng/ml: 50,000 IU/every 2 weeks for 4 weeks.
  Arms: 50,000 IU Vitamin D3

SUMMARY:
Primary hyperparathyroidism (PHPT) is a common disease that occurs in 1 in 10,000 people every year. In the presence of this condition, the parathyroid glands produce excessive amounts of parathyroid hormone (PTH), which regulates calcium levels. The high levels of parathyroid hormone remove too much calcium from bones, and then deposit the excess calcium in the blood, which is then filtered into the urine by the kidneys. Bone health is threatened by excess calcium loss which weakens bone structure. Other affected organs include the skeleton (calcium loss leads to a "weakening" of the skeleton), and the kidneys (high blood calcium can lead to kidney stones).

It is now evident that the majority of patients with even mild Primary Hyperparathyroidism are vitamin D deficient. In 2009, new international guidelines for the management of asymptomatic PHPT direct physicians to measure 25-hydroxyvitamin D (D3 or 25-OHD) in all patients, and to replete the reserve of vitamin D when the level is low (< 20 ng/ml). However, no recommendations for vitamin D repletion are given, because of limited data regarding the effects of vitamin D repletion, appropriate dosing and safety. Therefore, there is an urgent need for data upon which to base such recommendations, as well as are data on the effects of such treatment upon bones.

Subjects with low vitamin D3 levels will be selected for this trial. They will be given enough vitamin D3 to raise their low blood levels from a low to a normal range. The assessments in this study, including the quadruple label bone biopsy, will allow us to document the short term effects of administering vitamin D3 on changes in bone.

All participants enrolled in this trial will be vitamin D3 deficient. Participants will take an antibiotic (tetracycline) 4 times a day to mark the starting point from which bone changes will be assessed. After 3 days of tetracycline, a 12 week course of vitamin D3 or placebo will be initiated. Six of 7 participants will receive the study drug (active vitamin D3), while 1 in 7 will receive a placebo (sugar pill). Ten weeks later, another 3-day course of tetracycline will be given. At the end of 12 weeks, a bone biopsy will be done. A small piece of bone (about the size of a pencil eraser) will be removed from the hip (iliac crest). The bone will be analyzed to determine the effect of vitamin D3 on primary hyperparathyroidism.

There will be 4 study visits: Screening, Baseline, Week 8, and Week 12 when the bone biopsy will be performed.

Study Procedures:

Medical and Social History

Blood tests (drawn at the study center and local Quest Lab)

24-Hour urine collection for calcium and creatinine excretion

Abdominal X-ray (to assess for kidney stones)

Transiliac crest Bone Biopsy

ELIGIBILITY:
Inclusion Criteria:

1. Females and males >= 45 years of age
2. PHPT, defined as elevated PTH with elevated serum calcium
3. Screening 25-OHD <= 20 ng/ml

Exclusion Criteria:

1. Pre-menopausal
2. Serum calcium is >11.5mg/dl.
3. Urinary calcium is >350 mg/dl.
4. Active nephrolithiasis
5. Nephocalcinosis
6. Known sensitivity to tetracycline (Sumycin)
7. Familial history of hyperparathyroid syndromes
8. Bisphosphonate use within past 2 years.
9. Current use of Prolia.
10. Current use of Cinacalcet.
11. Currently using Cimetidine.
12. Currently use Colestipol.
13. Currently using Orlistat.
14. Current or past malignancy, except cured basal or squamous cell skin carcinoma or other cancers that have not recurred for at least five years.
15. Current tuberculosis, or history of Sarcoidosis, HIV/AIDS, chronic kidney disease (serum creatinine >= 1.5), liver disease, Crohn's Disease, Celiac Disease, or gastric bypass

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Bone Formation Rate (BFR) | 12 Weeks
  A between group (vitamin D3 vs. placebo) comparison of BFR will be performed at three surfaces, cancellous, intra- and endo-cortical.

CONTACTS AND LOCATIONS:
Overall Officials: Shonni J. Silverberg, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States